CLINICAL TRIAL: NCT04678544
Title: A Randomized Controlled Trial to Evaluate Effectiveness of Cooling Cap to Prevent Permanent Chemotherapy-induced Alopecia Among Breast Cancer Patients
Brief Title: Cooling Cap Trial to Prevent Permanent Chemotherapy-induced Alopecia in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Paxman (Unknown)
Responsible Party: Principal Investigator, Jin Seok Ahn, MD, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PAXMAN
Record Dates: First submitted 2020-11-24; First posted 2020-12-22 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Neoplasm, Breast
Keywords: Scalp cooling system; Randomized controlled trial; Permanent-Chemotherapy-Induced Alopecia; Chemotherapy-Induced Alopecia
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial, Single center
Who Masked: Outcomes Assessor
Masking Description: There will be no blindness of physician and patients. However, statisticians who will analyze the data will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): Before the chemotherapy, patients in intervention group will use cooling cap 30 minutes before chemotherapy. Once chemotherapy drug be ready, patients will receive chemotherapy. After the chemotherapy, patients go to the cooling cap area (room) and wear the cooling cap additional 20 minute for Taxane and 90 minute for other drugs, respectively.
  Interventions: Device: Scalp cooling system 2
- Controlled Group (No Intervention): chemotherapy with usual care

INTERVENTIONS:
Device: Scalp cooling system 2 — The investigational device which will be used in this study is the Paxman Scalp Cooling System 2. This device is manufactured by: Paxman Coolers Limited. This is a free-standing, electrically-powered, mobile refrigeration unit which circulates a refrigerated liquid coolant, at a pre-set temperature and flow rate, through a cooling cap which is attached to, and covers, the top of the patient's head. The Paxman Scalp Cooling System is intended to be used for scalp cooling of patients who are receiving chemotherapy for the treatment of solid tumors, in order to reduce the risk of chemotherapy-induced alopecia.
  After the RCT, 34 patients who were expected to receive 4, 6, or 8 cycles of chemotherapy with an anthracycline regimen were further enrolled in the intervention group as a single-arm trial.
  Arms: Intervention Group

SUMMARY:
This study aims to examine whether the PSCS2 is effective in reducing chemotherapy-induced alopecia in women with breast cancer undergoing neoadjuvant or adjuvant chemotherapy. Female adults who are newly diagnosed with stage 1-3 breast cancer and expected to receive Adriamycin or/Taxane will participate in the study. The study design is an open-label, randomized controlled trial. The patients will be randomly assigned to intervention or control groups. Intervention patients will have applied scalp cooling during 4 or 6 cycles of their chemotherapy. The primary endpoint is the effectiveness of the PSCS2 for reducing permanent chemotherapy-induced alopecia. Secondary endpoints include chemotherapy-induced alopecia, distress due to chemotherapy-induced alopecia, quality of life, and patient-reported alopecia-related side effects.

After the RCT, only patients who were expected to receive 4, 6, or 8 cycles of chemotherapy with an anthracycline regimen were further enrolled in the intervention group as a single-arm trial.

DETAILED DESCRIPTION:
Adjuvant chemotherapy decreases the risk of recurrence. However, it has distressing side effects, including alopecia. Chemotherapy-induced alopecia (CIA) is a common and distressing side effect of many chemotherapy drugs. In a previous study, more than half of the breast cancer patients experienced higher distress due to CIA during cancer treatment, and this distress was strongly associated with negative body image, overall health status, and psychosocial well-being. Recently scalp cooling has been known to be one of the effective options for hair loss prevention. However, there was little information regarding the effect on the prevention of permanent CIA(PCIA). This study aims to examine the impact of scalp cooling on the prevention of PCIA as well as CIA.

Female adults who are newly diagnosed with stage 1-3 breast cancer and aged less than 70 years will be screened for a plan of undergoing Adriamycin or/and Taxane regimen as neoadjuvant or adjuvant chemotherapy. Eligible patients will be randomly assigned to intervention or control groups (2:1 ratio). Patients in the intervention group will have applied scalp cooling during 4 or 6 cycles of their chemotherapy whereas participants in the control group will be observed.

The objective of the study is to examine whether the Paxman scalp cooling system is effective in reducing PCIA in women with breast cancer undergoing neoadjuvant or adjuvant chemotherapy. In addition, the impact of Paxman scalp cooling on the prevention of CIA, alopecia-related distress, quality of life, and patient-reported alopecia-related side effects will also be explored.

After the RCT, only patients who were expected to receive 4, 6, or 8 cycles of chemotherapy with an anthracycline regimen were further enrolled in the intervention group as a single-arm trial.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer, stage I-III
* Expected to receive 4 or 6 cycles of Adriamycin or Taxance of chemotherapy regimen as neoadjuvant or adjuvant chemotherapy with curative intent (e.g., AC, TC, or TCHP)
* For the additional single arm, patients who expected to receive 4, 6, or 8 cycles of Adriamycin or Taxance chemotherapy regimen as neoadjuvant or adjuvant chemotherapy with curative intent (e.g., AC, TC, TCHP, or AC+T).

Exclusion Criteria:

* Any other concurrent malignancy including hematological malignancies
* Elevated liver enzymes or bilirubin defined as 3 times the upper limits of normal
* Serum Albumin < 3.0
* Subjects who are underweight (defined as a BMI < 17.5)
* Subjects who have had previous chemotherapy exposure
* Subjects with cold agglutinin disease or cold urticarial
* Subject who had thyroid disease, diabetes or cardiac disease
* Subject who had auto-immune disease
* History of treatment due to alopecia
* Subject who had scalp disease

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Permanent chemotherapy-induced alopecia | 6 months (±2 months) after completion of chemotherapy and intervention
  Permanent chemotherapy-induced alopecia is defined as hair density or thickness less than two standard deviations (SDs) compared to the baseline mean (before chemotherapy) at 6 months (±2 months) after completion of chemotherapy. Hair density and thickness will be measured by using Folliscope 5.0, LeadM.

SECONDARY OUTCOMES:
Hair density and thickness during and after chemotherapy | Baseline, at the beginning (1st day) of the 2nd cycle (each cycle is 21days), 1month (±2 weeks) after completion of chemotherapy and intervention
  Hair density and thickness will be measured by using Folliscope 5.0, LeadM between 1st and 2nd intervention and at 1st clinical visit after chemotherapy compared to the baseline mean (before chemotherapy).
Distress due to chemotherapy-induced alopecia | Baseline, at the beginning (1st day) of the 2nd cycle (each cycle is 21days), 1month (±2 weeks) after completion of chemotherapy and intervention
  Chemotherapy-Induced Alopecia Distress Scale (CADS) will be used to demonstrate that the PSCS is effective in reducing distress due to chemotherapy-induced alopecia in woman with breast cancer undergoing neoadjuvant or adjuvant chemotherapy
Quality of life (cancer related quality of life) | Baseline, at the beginning (1st day) of the 2nd cycle (each cycle is 21days), 1month (±2 weeks) after completion of chemotherapy and intervention
  Quality of life will be measured using EORTC QLQ-C30. The QLQ-C30 is a cancer health-related quality-of-life questionnaire that has been widely used in clinical trials and investigations using patient reported outcome for individual patient management. It use a "past week" recall period. Raw scores are linearly converted to a 0-100 scale with higher scores reflecting higher levels of Quality of life.
Breast cancer related quality of life | Baseline, at the beginning (1st day) of the 2nd cycle (each cycle is 21days), 1month (±2 weeks) after completion of chemotherapy and intervention
  Quality of life will be measured using EORTC QLQ-BR23. The BR23 is a breast cancer specific module to measure health-related quality-of-life . It use a "past week" recall period. Raw scores are linearly converted to a 0-100 scale with higher scores reflecting higher levels of Quality of life.
Patients reported outcomes | Baseline, at the beginning (1st day) of the 2nd cycle (each cycle is 21days), 1month (±2 weeks) after completion of chemotherapy and intervention, and 6 months (±2 months) after completion of chemotherapy and intervention
  Self-reported hair loss will be assessed by using Korean version of PRO-CTCAE.
Global photographs | Baseline, at the beginning (1st day) of the 2nd cycle (each cycle is 21days), 1month (±2 weeks) after completion of chemotherapy and intervention, and 6 months (±2 months) after completion of chemotherapy and intervention
  Pictures to be focused on head/hair, which means shorter distance between the equipment and the subject by using Canon EOS 70D.

OTHER OUTCOMES:
Side effect | At the beginning (1st day) of the 2nd cycle (each cycle is 21days), At the beginning of 3rd cycle of chemotherapy, At the beginning of 4th cycle of chemotherapy, At the beginning of 5th cycle of chemotherapy, and , At the beginning 6th of chemotherapy
  Potential side-effect including discomfort due to the cold, headache, dizziness or vomiting.
Willingness to pay | At the beginning (1st day) of the 2nd cycle (each cycle is 21days), 1month (±2 weeks) after completion of chemotherapy, and 6 months (±2 months) after completion of chemotherapy
  Willingness to pay to use scalp cooling by self-developed questionnaire.
Effort for managing hair | Baseline, at the beginning (1st day) of the 2nd cycle (each cycle is 21days), 1month (±2 weeks) after completion of chemotherapy and intervention, and 6 months (±2 months) after completion of chemotherapy
  Usual care for hair and scalp, type of shampoo, wig
Characteristic of participants | Smoking, drinking, medication and exposure-time to sunlight at baseline, at the beginning (1st day) of the 2nd cycle (each cycle is 21days), and 6m (±2m) after completion of chemotherapy, the others at only baseline
  Demographic information including age, education, marital status, working status, income, smoking and drinking history, medication, exposure-time to sunlight and co-morbidities

CONTACTS AND LOCATIONS:
Overall Officials: Jin Seok Ahn, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Ilwon-ro 81, Gangnam-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The protocol summary, and informed consent form will be made available on clinicaltrials.gov when required.
  Requests for study protocol and informed consent form can be shared after starting recruit. Requests for deidentified individual participant data can be made beginning 24 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: jinseok.ahn@samsung.com or jcho@skku.edu
Supporting Information: Study Protocol, ICF
Time Frame: Requests for study protocol and informed consent form can be shared after starting recruit.
  Requests for deidentified individual participant data can be made beginning 24 months after publication and for up to 36 months post publication.
Access Criteria: People who send a request e-mail and be received confirmation from : jinseok.ahn@samsung.com or jcho@skku.edu

REFERENCES:
- [Background] McGarvey EL, Baum LD, Pinkerton RC, Rogers LM. Psychological sequelae and alopecia among women with cancer. Cancer Pract. 2001 Nov-Dec;9(6):283-9. doi: 10.1046/j.1523-5394.2001.96007.x. PMID 11879330
- [Background] Batchelor D. Hair and cancer chemotherapy: consequences and nursing care--a literature study. Eur J Cancer Care (Engl). 2001 Sep;10(3):147-63. doi: 10.1046/j.1365-2354.2001.00272.x. PMID 11829374
- [Background] Choi EK, Kim IR, Chang O, Kang D, Nam SJ, Lee JE, Lee SK, Im YH, Park YH, Yang JH, Cho J. Impact of chemotherapy-induced alopecia distress on body image, psychosocial well-being, and depression in breast cancer patients. Psychooncology. 2014 Oct;23(10):1103-10. doi: 10.1002/pon.3531. Epub 2014 Mar 24. PMID 24664939
- [Background] Kim IR, Cho J, Choi EK, Kwon IG, Sung YH, Lee JE, Nam SJ, Yang JH. Perception, attitudes, preparedness and experience of chemotherapy-induced alopecia among breast cancer patients: a qualitative study. Asian Pac J Cancer Prev. 2012;13(4):1383-8. doi: 10.7314/apjcp.2012.13.4.1383. PMID 22799336
- [Background] Cho J, Choi EK, Kim IR, Im YH, Park YH, Lee S, Lee JE, Yang JH, Nam SJ. Development and validation of Chemotherapy-induced Alopecia Distress Scale (CADS) for breast cancer patients. Ann Oncol. 2014 Feb;25(2):346-51. doi: 10.1093/annonc/mdt476. Epub 2013 Dec 29. PMID 24379161
- [Background] Dunnill CJ, Al-Tameemi W, Collett A, Haslam IS, Georgopoulos NT. A Clinical and Biological Guide for Understanding Chemotherapy-Induced Alopecia and Its Prevention. Oncologist. 2018 Jan;23(1):84-96. doi: 10.1634/theoncologist.2017-0263. Epub 2017 Sep 26. PMID 28951499
- [Background] Breed WP. What is wrong with the 30-year-old practice of scalp cooling for the prevention of chemotherapy-induced hair loss? Support Care Cancer. 2004 Jan;12(1):3-5. doi: 10.1007/s00520-003-0551-8. Epub 2003 Nov 13. PMID 14615930
- [Background] Rugo HS, Melin SA, Voigt J. Scalp cooling with adjuvant/neoadjuvant chemotherapy for breast cancer and the risk of scalp metastases: systematic review and meta-analysis. Breast Cancer Res Treat. 2017 Jun;163(2):199-205. doi: 10.1007/s10549-017-4185-9. Epub 2017 Mar 8. PMID 28275922
- [Background] Nangia J, Wang T, Osborne C, Niravath P, Otte K, Papish S, Holmes F, Abraham J, Lacouture M, Courtright J, Paxman R, Rude M, Hilsenbeck S, Osborne CK, Rimawi M. Effect of a Scalp Cooling Device on Alopecia in Women Undergoing Chemotherapy for Breast Cancer: The SCALP Randomized Clinical Trial. JAMA. 2017 Feb 14;317(6):596-605. doi: 10.1001/jama.2016.20939. PMID 28196254
- [Background] Rugo HS, Klein P, Melin SA, Hurvitz SA, Melisko ME, Moore A, Park G, Mitchel J, Bageman E, D'Agostino RB Jr, Ver Hoeve ES, Esserman L, Cigler T. Association Between Use of a Scalp Cooling Device and Alopecia After Chemotherapy for Breast Cancer. JAMA. 2017 Feb 14;317(6):606-614. doi: 10.1001/jama.2016.21038. PMID 28196257
- [Background] Kluger N, Jacot W, Frouin E, Rigau V, Poujol S, Dereure O, Guillot B, Romieu G, Bessis D. Permanent scalp alopecia related to breast cancer chemotherapy by sequential fluorouracil/epirubicin/cyclophosphamide (FEC) and docetaxel: a prospective study of 20 patients. Ann Oncol. 2012 Nov;23(11):2879-2884. doi: 10.1093/annonc/mds095. Epub 2012 May 9. PMID 22571858
- [Background] Kang D, Kim IR, Im YH, Park YH, Ahn JS, Lee JE, Nam SJ, Park H, Kim E, Lee HK, Lee DY, Cho J. Quantitative changes in skin composition parameters due to chemotherapy in breast cancer patients: a cohort study. Breast Cancer Res Treat. 2015 Aug;152(3):675-82. doi: 10.1007/s10549-015-3502-4. Epub 2015 Jul 22. PMID 26198993
- [Background] Kang D, Kim IR, Choi EK, Im YH, Park YH, Ahn JS, Lee JE, Nam SJ, Lee HK, Park JH, Lee DY, Lacouture ME, Guallar E, Cho J. Permanent Chemotherapy-Induced Alopecia in Patients with Breast Cancer: A 3-Year Prospective Cohort Study. Oncologist. 2019 Mar;24(3):414-420. doi: 10.1634/theoncologist.2018-0184. Epub 2018 Aug 17. PMID 30120165
- [Background] Kim SN, Lee SY, Choi MH, Joo KM, Kim SH, Koh JS, Park WS. Characteristic features of ageing in Korean women's hair and scalp. Br J Dermatol. 2013 Jun;168(6):1215-23. doi: 10.1111/bjd.12185. PMID 23278260
- [Background] Janssen FP, Rajan V, Steenbergen W, van Leeuwen GM, van Steenhoven AA. The relationship between local scalp skin temperature and cutaneous perfusion during scalp cooling. Physiol Meas. 2007 Aug;28(8):829-39. doi: 10.1088/0967-3334/28/8/006. Epub 2007 Jul 6. PMID 17664675
- [Background] Bulow J, Friberg L, Gaardsting O, Hansen M. Frontal subcutaneous blood flow, and epi- and subcutaneous temperatures during scalp cooling in normal man. Scand J Clin Lab Invest. 1985 Oct;45(6):505-8. doi: 10.3109/00365518509155250. PMID 4070952
- [Background] Lane P, Vichi P, Bain DL, Tritton TR. Temperature dependence studies of adriamycin uptake and cytotoxicity. Cancer Res. 1987 Aug 1;47(15):4038-42. PMID 3607749
- [Background] Gregory RP, Cooke T, Middleton J, Buchanan RB, Williams CJ. Prevention of doxorubicin-induced alopedia by scalp hypothermia: relation to degree of cooling. Br Med J (Clin Res Ed). 1982 Jun 5;284(6330):1674. doi: 10.1136/bmj.284.6330.1674. No abstract available. PMID 6805650
- [Background] Komen MMC, Smorenburg CH, Nortier JWR, van der Ploeg T, van den Hurk CJG, van der Hoeven JJM. Results of scalp cooling during anthracycline containing chemotherapy depend on scalp skin temperature. Breast. 2016 Dec;30:105-110. doi: 10.1016/j.breast.2016.09.007. Epub 2016 Sep 28. PMID 27689316
- [Background] van den Hurk CJ, Peerbooms M, van de Poll-Franse LV, Nortier JW, Coebergh JW, Breed WP. Scalp cooling for hair preservation and associated characteristics in 1411 chemotherapy patients - results of the Dutch Scalp Cooling Registry. Acta Oncol. 2012 Apr;51(4):497-504. doi: 10.3109/0284186X.2012.658966. Epub 2012 Feb 6. PMID 22304489
- [Background] Komen MM, Breed WP, Smorenburg CH, van der Ploeg T, Goey SH, van der Hoeven JJ, Nortier JW, van den Hurk CJ. Results of 20- versus 45-min post-infusion scalp cooling time in the prevention of docetaxel-induced alopecia. Support Care Cancer. 2016 Jun;24(6):2735-41. doi: 10.1007/s00520-016-3084-7. Epub 2016 Jan 25. PMID 26805558
- [Background] Kang D, Kim IR, Park YH, Im YH, Zhao D, Guallar E, Ahn JS, Cho J. Impact of a topical lotion, CG428, on permanent chemotherapy-induced alopecia in breast cancer survivors: a pilot randomized double-blind controlled clinical trial (VOLUME RCT). Support Care Cancer. 2020 Apr;28(4):1829-1837. doi: 10.1007/s00520-019-04982-z. Epub 2019 Jul 23. PMID 31338640
- [Derived] Kang D, Cho J, Zhao D, Kim J, Kim N, Kim H, Kim S, Kim JY, Park YH, Im YH, Guallar E, Ahn JS. Scalp Cooling in Preventing Persistent Chemotherapy-Induced Alopecia: A Randomized Controlled Trial. J Clin Oncol. 2024 Sep 10;42(26):3115-3122. doi: 10.1200/JCO.23.02374. Epub 2024 Jun 6. PMID 38843479